CLINICAL TRIAL: NCT01612936
Title: T Cell Effector and Regulatory Mechanisms in Asthma
Acronym: MGH-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew D. Luster, M.D.,Ph.D. (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Andrew D. Luster, M.D.,Ph.D., Chief, Division of Rheumatology, Allergy, and Immunology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012P000705; 1U19AI095261 (NIH)
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Asthma; Allergies
Keywords: Asthma; Allergic; Inflammation; Constriction; Airway; Challenge; Chemokines
MeSH Terms: conditions — Asthma; Hypersensitivity; Inflammation; Constriction, Pathologic | interventions — Bronchoscopy; Ventilation; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allergic asthmatic, allergic nonasthmatic (Experimental): Adults who are allergic asthmatics or allergic non-asthmatics will receive segmental allergen challenge to the lung
  Interventions: Biological: Bronchoscopy, Segmental Allergen Challenge and Broncheoalveolar Lavage; Procedure: PET-CT imaging(13NN perfusion/ventilation, 18FDG inflammation, and CT imaging)

INTERVENTIONS:
Biological: Bronchoscopy, Segmental Allergen Challenge and Broncheoalveolar Lavage — On the day of the first bronchoscopy,BAL will first be performed in the lingula without instillation of diluent or allergen.Then, a 2-ml aliquot of isotonic diluent is instilled into the right upper lobe. Then, the procedure will be repeated in the right middle lobe with instillation of 2-ml of standardized cat or mite allergen solution.A "test dose" concentration of allergen is administered first consisting of 2 ml of allergen at 1/10th(Cat,D.farinae) or 1/30th(D. pteronyssinus) the threshold concentration.If on visual inspection through the bronchoscope, there is no evidence of mucosal inflammation after two minutes, a second segmental allergen challenge will be done in the right middle lobe using 2-ml of full-dose allergen at the threshold concentration(Cat,D.farinae) or 1/3th the threshold concentration(D.pteronyssinus).This dose will be predetermined by quantitative skin prick testing.A second bronchoscopy is performed 24 hours after delivery of allergen extract and diluent.
  Other Names: One of 3 Standardized allergen extracts will be used:; 1)Cat hair; 2)Dust Mite Dermatophagoides farinae; 3)Dust Mite Dermatophagoides pteronyssinus; Phenolized saline diluent will also be used in this study.; All will be purchased from Greer Laboratories, Lenoir, NC.
Procedure: PET-CT imaging(13NN perfusion/ventilation, 18FDG inflammation, and CT imaging) — Imaging is first performed the evening prior to the 1st bronchoscopy.An IV catheter is placed.An attenuation correction is performed to remove image distortion using a chest CT volumetric scan.Subjects are instructed to exhale to the same mean lung volume of the CT scan and hold their breath for 20sec.Simultaneous with apnea,13NNsaline is injected IV and a series of PET scans is acquired.Then subjects resume breathing, matching their previous respiratory rate and tidal volume.After 3 min,within an interval of 1 min,spirometry and 2 deep inhalations are performed,followed by 1 min of washout. For the second imaging visit, which will occur 24 hour later, the imaging sequence will be repeated as described above, but will also include 18FDG infusion.At least 30 minutes after the 13NN injection,10mCi of 18FDG is infused. Then, images are collected over a 75 minutes.Venous blood is sampled at 5 different time points over a 40-45 minute time window to determine plasma radioactive levels.
  Other Names: 13N-N2 saline; 18F-FDG, 0.019 mSv/MBq

SUMMARY:
The specific hypothesis for this study is that there are fundamental differences in T effector and T regulatory cell responses in the lung to allergens in allergic asthma (AA) when compared to allergic nonasthmatics (ANA) that account for the difference in clinical responses. We will address this by comparing T cell responses in AA versus ANA subjects. These experiments will correlate T cell responses with measures of airway physiology using state-of-the art lung imaging and examine mechanisms controlling T cell activation in the airways of AA and the function of airway T regulatory cells during AA.

DETAILED DESCRIPTION:
Despite advances in medications, allergic diseases, including allergic asthma, continue to rise in prevalence. For this reason, there is a need for a better understanding of the mechanisms of allergic diseases and novel insights into modulating allergic inflammation. CD4+ Th2-type lymphocytes seems to be central to the pathogenesis of allergic disease, as the levels of these cells and Th2 cytokines (IL-4, IL-5 and IL-13) are elevated in the airways of allergic asthma patients. The unifying hypothesis of this project is that understanding the mechanisms that determine the critical balance of effector and regulatory allergen-specific T cell activity in asthma will lead to new approaches for inducing allergen-specific tolerance and new therapeutic strategies for asthma.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Allergic Asthma (AA subjects):

1. All subjects will have a baseline FEV1 no less than 75 % of the predicted value after bronchodilator administration.
2. All subjects will have both a clinical history of allergic symptoms to cat or dust mite allergen and a positive allergen prick test (3 mm diameter greater than diluent control)
3. Life-long absence of cigarette smoking (lifetime total of < 5 pack-years and none in 5 years).
4. Willing and able to give informed consent.
5. Expressed the desire to participate in an interview with the principal investigator.
6. Age between 18 and 50 years.
7. A methacholine PC20 < 16 mg/ml.
8. Asthma of severity defined as: requiring no more than step 3 therapy (NHLBI Guidelines, 2007 EPR-3, http://www.nhlbi.nih.gov/guidelines/asthma/asthgdln.pdf), well-controlled and having a validated asthma control test (ACT) score of > 19 for one month prior to the screening visit, and able to tolerate a 2 week stoppage of inhaled corticosteroids prior to Visit 2.

Allergic Nonasthmatic Subjects (ANA subjects):

1. ANA subjects will have a history of at least one of the following: (a) allergic rhinitis (with one or more of the following symptoms: nasal congestion, sneezing, runny nose, postnasal drainage), (b) allergic conjunctivitis (ocular itching, tearing and/or swelling) or (c) contact allergy associated with cat dander or dust mite and a positive allergy test to the same allergen.
2. All subjects will have a baseline FEV1 and FVC determined at the characterization visit that is no less than 90 % of the predicted value before bronchodilator administration.
3. All subjects will have a positive allergy skin prick test to cat dander or dust mite allergen.
4. All subjects will be in good general health.
5. Life-long absence of cigarette smoking (lifetime total of < 5 pack-years and none in 5 years).
6. Willing and able to give informed consent.
7. Expressed the desire to participate in an interview with the principal investigator.
8. Age between 18 and 50 years.

Exclusion Criteria:

Subjects with Allergic Asthma (AA subjects):

1. Women of childbearing potential who are pregnant (based on urine beta-HCG or STAT quantitative serum hCG testing), are sexually active and not using contraception, are seeking to become pregnant, or who are nursing.
2. The presence of spontaneous asthmatic episode or clinical evidence of upper respiratory tract infection within the previous 6 weeks.
3. Participation in a research study involving a drug or biologic during the 30 days prior to the study.
4. Intolerance to albuterol, atropine, lidocaine, fentanyl, or midazolam.
5. Antihistamines within 7 days of the screening visit.
6. Presence of diabetes mellitus, congestive heart failure, ventricular arrhythmias, history of a cerebrovascular accident, renal failure, history of anaphylaxis, or cirrhosis.
7. Use of systemic steroids, increased use of inhaled steroids, beta blockers and MAO inhibitors or a visit for an asthma exacerbation within 1 month of the screening visit.
8. Antibiotic use for respiratory disease within 1 month of the characterization visit or a respiratory tract infection within 6 weeks of the bronchoscopy visits.
9. A history of asthma-related respiratory failure requiring intubation.
10. Quantitative skin-prick test positive reaction down to an allergen concentration of 0.056 BAU or AU/ml.
11. Subjects with a high possibility of poor compliance with the study.
12. Have a history of cigarette smoking within the past 5 years or > 5 pack years total.
13. Having second-hand cigarette smoke exposure or indoor furry pets except in the case of dog, if the subject is not allergic to the dog and the subject has a negative skin test to dog.
14. Other lung diseases, such as sarcoidosis, bronchiectasis or active lung infection.
15. Use of Xolair (omalizumab - anti-IgE monoclonal antibody) for 6 months.
16. Immunotherapy with cat or dust mite extract now or in the past.
17. Use of prophylactic aspirin for cardiovascular disease
18. Non-English speakers

Allergic Nonasthmatic Subjects (ANA subjects):

1. A history of asthma.
2. Exclusion criteria #1, 3-8 and 10- 18 from (AA) above.
3. A methacholine PC20 < 16 mg/ml.

Additional exclusion Criteria Specific to PET Imaging:

1. Anyone unable to lay flat on the scanner table for imaging.
2. We will exclude severely and morbidly obese subjects (BMI> 32) because of the poor quality of images that can be obtained and weight restrictions on the scanner.
3. Those with a diffusing capacity < 80% predicted (if known),
4. Subjects with known exposure to agents that are associated with pulmonary disease (i.e. asbestos, silica)
5. Subjects who have had any research related radiation exposure greater than 15 mSv within the past year will be excluded.
6. Individuals with known allergy or hypersensitivity to FDG will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Differences in airway physiology and airway constriction | 24 hours
  The primary endpoints are differences in airway physiology and airway constriction following segmental allergen challenge (SAC) in AA and ANA subjects using positron emission tomography (PET) in combination with high-resolution computed tomography (HRCT)

SECONDARY OUTCOMES:
Differences in BAL inflammatory mediator release | 24 hours
  We will assess each BAL for inflammation and inflammatory mediator release. A pre-challenge BAL is obtained to insure the subject does not have baseline inflammation prior to the allergen challenge. The diluent challenged segment is used to control for effects of bronchoscopy and instillation of fluid in the lung. Analysis of the allergen challenged segment is done to confirm that allergen exposure led to airway inflammation, and allows us to correlate changes in airway physiology to inflammation in the allergen exposed segment.
Differences in cellular analysis of BAL | 24 hours
  A differential is calculated for each sample by counting at least 200 cells using morphology and staining characteristics to separate them into macrophages, lymphocytes, eosinophils, and neutrophils, allowing us to calculate the number and percentage of each cell type in the BAL. The cells are also stained for a panel of cell surface markers and intracytoplasmic proteins and analyzed by flow cytometry. This analysis will allow us to ensure that each subject responded to allergen challenge response with appropriate eosinophil and T cell recruitment into the BAL.
Differences in BAL inflammatory protein levels | 24 hours
  BAL fluid will be concentrated 10-fold using a Centricon filter (Millipore) with a 3,000 MW cutoff. We have found that assaying for cytokines is more reliable when the BAL is concentrated 10-fold since BAL is diluted ~100-fold by the procedure.Concentrations of a panel of 42 different cytokines, chemokines, and growth factors are measured using a LINCOplex human cytokine-chemokine kit as per manufacturer's guidelines (Millipore) and read on a Luminex 100 (Luminex Corporation). Results are analyzed using Beadview software (UpstateCell Signaling Solutions).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Luster, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States